CLINICAL TRIAL: NCT06617260
Title: Longitudinal FolloW-up of Antimicrobial Resistance From Perinatal Acquisition (LWAPA): A SHARE Study ASSESSING AND PREVENTING Antimicrobial Resistance in the Perinatal Period
Acronym: LWAPA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ebbing Lautenbach, Professor of Medicine, University of Pennsylvania
Other Study IDs: 855283; Antimicrobial resistance(AMR), (Other: the U.S. Centers for Disease Control & Prevention)
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Drug Resistance, Microbial
Keywords: Antimicrobial

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Rectovaginal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates and mothers: Pre-partum mothers will be eligible for recruitment if they have been admitted to the pre-partum ward (2F) at PMH. This includes mothers with:
  * Pre-term labor (24-36 weeks gestation)
  * Pre-eclampsia
  * Post-dates (>41 weeks gestation) The rationale for recruiting these mothers is that there is a high probability of having a baby who will ultimately be admitted to the NNU

SUMMARY:
In 2022, in collaboration between the Botswana Ministry of Health (MOH), the U.S. Centers for Disease Control & Prevention, and the Botswana-UPenn Partnership (BUP), a program was launched called, "Surveillance of Healthcare-associated infections & Antimicrobial Resistance", or "SHARE". The aims of SHARE are to 1) enhance laboratory capacity to detect emerging AMR patterns; 2) strengthen hospital epidemiology programs, leveraging data to prevent, detect, and contain emerging AMR threats; 3) deploy study teams to answer critical public health surveillance questions, and 4) to build a national network of hospital infection prevention and control (IPC) resources to prevent, detect, and contain emerging infectious disease threats.

DETAILED DESCRIPTION:
The Longitudinal FolloW-up of Antimicrobial Resistance from Perinatal Acquisition (LWAPA) study will assess the extent of perinatally-acquired MDROs and GBS, exploring factors influencing both maternal and neonatal colonization and better understanding the long-term outcomes in families affected by MDRO colonization.

By collecting samples at critical time points (e.g. during labour, after delivery, sequentially in the hospital, and then 3, 6, 9, and 12 months of age, the LWAPA study aims to identify modifiable factors influencing colonization risk. The results from this study can help inform and operationalize infection prevention measures which are poised to reduce the incidence of healthcare-associated infections and other poor health outcomes.

In Setswana, 'lwapa' means 'home' or 'family', which captures how this study aims to understand healthcare-associated AMR is impacting households and communities.

ELIGIBILITY:
Inclusion Criteria:

Pre-partum mothers will be eligible for recruitment if they have been admitted to the pre-partum ward (2F) at PMH. This includes mothers with:

* Pre-term labor (24-36 weeks gestation)
* Pre-eclampsia
* Post-dates (>41 weeks gestation)-

Exclusion Criteria:

Mothers/babies who have been admitted for more than 96 hours will be excluded

Min Age: 36 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pre partum mothers
Study Population: Pre-partum mothers will be eligible for recruitment if they have been admitted to the pre-partum ward (2F) at PMH. This includes mothers with:
  * Pre-term labor (24-36 weeks gestation)
  * Pre-eclampsia
  * Post-dates (>41 weeks gestation) The rationale for recruiting these mothers is that there is a high probability of having a baby who will ultimately be admitted to the NNU
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Longitudinal FolloW-up of Antimicrobial Resistance from Perinatal Acquisition | 12 months
  Ultimately, the goal of the LWAPA study is to better understand perinatal transmission of AMR in order to inform prevention measures

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana